CLINICAL TRIAL: NCT00609648
Title: Distance Psychology for Treating Dental Fear in Rural Communities
Brief Title: Computer Assisted Relaxation Learning for Dental Offices
Acronym: CARL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Sue Coldwell, Study Principal Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 30641-B; U54DE014254 (NIH); U01DE016750 (NIH); U01DE016752 (NIH)
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Dental Anxiety
Keywords: Dental Anxiety; Dental Phobia; Odontophobia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CARL (Experimental): CARL computer program
  Interventions: Behavioral: Computer Assisted Relaxation Learning
- Pamphlet (Active Comparator): Reassuring pamphlet about dental injections
  Interventions: Behavioral: Pamphlet

INTERVENTIONS:
Behavioral: Computer Assisted Relaxation Learning — A self-paced computer program for reducing dental injection fear.
  Arms: CARL
Behavioral: Pamphlet — A pamphlet reassuring patients about dental injections.
  Arms: Pamphlet

SUMMARY:
This is a randomized study in which two groups will be used to compare the effectiveness of a computerized psychological therapy compared to an information only control group (pamphlet) for reducing fear of dental injections.

DETAILED DESCRIPTION:
This is a randomized study in which two groups will be used to compare the effectiveness of a computerized psychological therapy compared to an information only control group (pamphlet) for reducing fear of dental injections. All patients (96 people with high fear of dental injections) will be tested to assess pre-existing dental fear levels prior to being assigned to study condition. Subsequently, patients in the active treatment group will complete computerized psychological therapy in 1 to 9 weekly 45-minute sessions. Subjects in the control condition will meet with a dental assistant once for approximately 15 minutes to go over a pamphlet. The pamphlet is based on written information developed by a commercial dental web site development company. Following the intervention or control procedures, patients will be reassessed for dental fear using computerized questionnaires. They will also be scheduled to receive a dental injection. Subjects' willingness to complete the dental injection and fear levels during the dental injection will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* High dental injection fear
* Age 18 and over
* Healthy with no untreated systemic conditions
* Able to read and write English

Exclusion Criteria:

* Heart murmur
* Known allergies to lidocaine or benzocaine
* Under 18 year old
* Untreated systemic conditions
* Currently receiving medication for anxiety

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2008-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Modified Interval Scale of Anxiety Response at dental injection appointment | One to two-weeks post-intervention/control

SECONDARY OUTCOMES:
Completion of the behavioral avoidance test | One to two-weeks post-intervention/control
Needle Survey | Immediately post-intervention/control
Modified Dental Anxiety Scale | Immediately post-intervention/control
Dental Fear Survey | Immediately post-intervention/control

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Coldwell, PhD, Principal Investigator — University of Washington
Locations (5):
- United States (5):
  - Dr. Gary Templeman, DDS, Corvallis, Oregon
  - Michael C Hazel, DMD, PC, West Linn, Oregon
  - Northwest Dental Fears Research, Bremerton, Washington
  - Valley View Health Center, Chehalis, Washington
  - Dental Fears Research Clinic, Seattle, Washington

REFERENCES:
- [Background] Coldwell SE, Getz T, Milgrom P, Prall CW, Spadafora A, Ramsay DS. CARL: a LabVIEW 3 computer program for conducting exposure therapy for the treatment of dental injection fear. Behav Res Ther. 1998 Apr;36(4):429-41. doi: 10.1016/s0005-7967(97)10038-9. PMID 9670603
- [Derived] Heaton LJ, Leroux BG, Ruff PA, Coldwell SE. Computerized dental injection fear treatment: a randomized clinical trial. J Dent Res. 2013 Jul;92(7 Suppl):37S-42S. doi: 10.1177/0022034513484330. Epub 2013 May 20. PMID 23690352